CLINICAL TRIAL: NCT07163104
Title: The Effects of Three Different Nonpharmacological Methods Used in Subcutaneous Application on Pain, Anxiety, and Fear Levels in Children With Oncology Diagnosis
Brief Title: The Effects of Nonpharmacological Methods Used in Subcutaneous Application on Pain, Anxiety, and Fear Levels in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zubeyde Ezgi Ercelik (Other)
Responsible Party: Sponsor-Investigator, Zubeyde Ezgi Ercelik, Assistant Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25/03
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Oncology
Keywords: Childhood cancer; Pain management; Anxiety; Invasive procedures; Subcutaneous injections; Nonpharmacological interventions; Nursing care; Pediatric oncology
MeSH Terms: conditions — Neoplasms; Agnosia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kaleidoscope (Experimental): After subcutaneous administration, children will rate their pain levels during and after the procedure with the Wong Baker Scale, their anxiety levels with the Children's State Anxiety Scale (CSA), and their fear levels with the Children's Fear Scale (CFS). A parent present with the child will observe the child's behavioral state during the procedure and will rate the child's fear level during and after the procedure with the CFS and their anxiety level with the CSA.
  Interventions: Behavioral: Kaleidoscope
- Buzzy (Experimental): For children in this group, a Buzzy device will be placed on the treatment area 60 seconds before the subcutaneous application begins, and cold and vibration will be applied. At the end of this period, the nurse will slide the Buzzy device approximately 3 cm above the treatment area, and the procedure will be performed. The Buzzy device will continue throughout the procedure, and once the procedure is complete, the Buzzy device will be removed. After subcutaneous administration, children will rate their pain levels during and after the procedure with the Wong Baker Scale, their anxiety levels with the Children's State Anxiety Scale (CSA), and their fear levels with the Children's Fear Scale (CFS). A parent present with the child will observe the child's behavioral state during the procedure and will rate the child's fear level during and after the procedure with the CFS and their anxiety level with the CSA.
  Interventions: Behavioral: Buzzy
- Cognitive behavioral intervention (Experimental): It consists of four components: procedural preparation and information, cognitive distraction, suggestions and caregiver education (cognitive components), and cognitive distraction and positive reinforcement (behavioral components).
  Interventions: Behavioral: Cognitive behavioral intervention

INTERVENTIONS:
Behavioral: Kaleidoscope — Immediately before the procedure, children will be given the opportunity to examine the kaleidoscope and asked what shapes they see. The kaleidoscope distraction will begin immediately before the immunotherapy procedure and continue throughout the procedure. Children will be asked detailed questions such as, "What shapes do you see in the picture? What colors are there? How many eyes do you see in the picture?", which the child can only accurately answer after careful examination. After the procedure, the kaleidoscope will be wiped with 70% alcohol and preserved by the researcher for the next session. A Zapp Flex Kaleidoscope (31.5 cm) will be used in this study.
  Arms: Kaleidoscope
Behavioral: Buzzy — The device contains a wing-shaped ice pack on the skin-contact portion. The ice pack is stored in a deep freezer and inserted into the device before application. After application, the ice pack is wiped with 70% alcohol and kept in the freezer until it freezes again. Cold application and vibration begin before the procedure and continue until the end. When vibration is applied, it reduces or eliminates pain by causing numbness, paresthesia, and anesthesia. Cold application reduces pain by slowing or blocking conduction in peripheral nerves. It also reduces pain by activating the gate-control mechanism, stimulating touch receptors, and increasing the release of endogenous opioids.
  Arms: Buzzy
Behavioral: Cognitive behavioral intervention — The researcher will suggest various distraction techniques (counting, singing, reading poetry, answering questions, etc.) to shift the child's focus during the procedure. The distraction technique chosen by the child will be used during the procedure. This method will be chosen during the preparation and briefing phases of the procedure. Cognitive behavioral intervention application will begin before subcutaneous application and will last 15-20 minutes, after which subcutaneous application will begin. After subcutaneous administration, children will rate their pain levels during and after the procedure with the Wong Baker Scale, their anxiety levels with the Children's State Anxiety Scale (CSA), and their fear levels with the Children's Fear Scale (CFS). A parent present with the child will observe the child's behavioral state during the procedure and will rate the child's fear level during and after the procedure with the CFS and their anxiety level with the CSA.
  Arms: Cognitive behavioral intervention

SUMMARY:
Childhood cancers are increasing globally and require long-term invasive treatments, particularly subcutaneous applications that often cause pain, swelling, and anxiety. Effective pain and anxiety management is essential, as early traumatic experiences may shape children's future pain responses. Nonpharmacological methods-classified as physical, cognitive, and behavioral-are widely used alongside pharmacological strategies due to their safety, cost-effectiveness, and ease of application. Although studies show these methods reduce pain and anxiety, there is still a need for high-quality research comparing multiple approaches across different age groups and procedures. This study aims to evaluate and compare the effectiveness of combined physical, cognitive, and behavioral interventions in managing pain, anxiety, and fear among children with oncological diagnoses undergoing invasive procedures.

DETAILED DESCRIPTION:
Childhood cancers have become an important public health problem due to their rapidly increasing incidence worldwide. Global and national data indicate not only a significant rise in childhood cancer cases but also show that countries' levels of development affect treatment success (Kutluk et al., 2023; WHO, 2024). Long-term treatment protocols, chemotherapy, and radiotherapy result in many invasive procedures in children, with subcutaneous applications being frequently used. Although subcutaneous administration has fewer systemic side effects compared to other methods, the likelihood of local and acute reactions remains high. The most common physical reactions experienced by children are pain, swelling, and redness at the injection site, while emotional reactions frequently include fear and anxiety (Arasi et al., 2018; Endaryanto & Nugraha, 2021; Mahler et al., 2020). From birth, children are exposed to many invasive procedures and experience pain and anxiety. McCaffery defined pain as "whatever the experiencing person says it is, existing whenever he says it does," emphasizing its subjective nature (McCaffery, 1968). Painful procedures encountered early in life, if not managed appropriately, may shape children's future pain responses and become a source of trauma (Birnie et al., 2019; Zieliński, Morawska-Kochman & Zatoński, 2020). Therefore, proper pain management during childhood is crucial in reducing the traumatic impact of painful experiences. This is particularly important for children undergoing repeated and long-term procedures such as immunotherapy, where pain and anxiety should be effectively managed during interventions (Ahmadpour et al., 2020).

The American Academy of Pediatrics (AAP) and the American Pain Society recommend alleviating pain and anxiety even during minor procedures. Effective and timely pain control during invasive medical procedures not only reduces immediate distress but also increases tolerance in subsequent procedures. The AAP highlighted the importance of pain management in patient care by defining pain as the "fifth vital sign" to raise awareness among healthcare professionals (AAP, 2022).

Pain and anxiety control requires a multidisciplinary team approach, with nurses playing a key role. Accurate identification, assessment, and management of children's pain are central to nursing care (Alotaibi et al., 2018). The American Society for Pain Management Nursing (ASPMN) emphasizes nurses' responsibility in ensuring pain control before, during, and after invasive procedures through both pharmacological and nonpharmacological methods. Multiple strategies exist to reduce pain and anxiety in pediatric invasive procedures. The use of nonpharmacological methods, either alone or in combination with pharmacological treatments, has increased in recent years due to their effectiveness in reducing pain, as well as their safety, ease of use, low cost, and time efficiency. Selection of nonpharmacological interventions should consider the child's cognitive capacity, age, culture, behavioral characteristics, coping skills, and type of pain (Addab et al., 2022; Erdoğan & Özdemir, 2021; Czech et al., 2021).

Nonpharmacological interventions in children are classified into physical, cognitive, and behavioral methods. In the literature, these methods have been applied during vaccinations, injections, blood draws, pre- and postoperative care, and dressing changes (Sivri et al., 2022; Topçu et al., 2022; Yılmaz & Şahiner, 2022). While existing studies show that nonpharmacological interventions are effective in reducing pain and anxiety during invasive procedures, further high-quality studies are needed to evaluate easily applicable approaches across different age groups. In this context, it is important to conduct research comparing the effectiveness of multiple nonpharmacological methods in controlling pain, anxiety, and fear in various pediatric procedures. This study aims to contribute to the literature by simultaneously applying and comparing three types of interventions-physical, cognitive, and behavioral-among children with oncological diagnoses to evaluate their effectiveness in pain and anxiety management.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-14 years,
* Have an oncological diagnosis,
* Have received at least one chemotherapy treatment before,
* And whose parents are willing to participate in the study will be included in the study.

Exclusion Criteria:

* Children with any visual, auditory, verbal, or cognitive impairment,
* Those in the terminal stages of their illness,
* Those with a history of sedative, analgesic, or narcotic use within 24 hours of admission,
* Those with a febrile illness or history of infection at the time of admission,
* Those with a score of 2 or higher on the Wong-Baker Pain Scale independent of the procedure (during the pre-procedure assessment),
* Those who do not complete the study will not be included in the study.

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Child Fear Scale and Child State Anxiety Scale | 5 minutes after the procedure
  This method is used to measure children's fear and anxiety. Children are shown pictures of five facial expressions, each scored between 0 and 4. A score of 0 indicates no fear or anxiety, while a score of 4 indicates the highest level of fear and anxiety. These are:
  * "0" represents a neutral expression (no anxiety)
  * "1" represents very little fear (very little anxiety)
  * "2" represents some fear (some anxiety)
  * "3" represents more fear (more anxiety)
  * "4" represents the highest level of fear (severe anxiety).
Wong-Baker Faces Pain Rating Scale | 5 minutes after the procedure
  Six facial expressions are scored from left to right, from 0 to 5 (0 = very happy/no pain, 5 = most severe pain). As the score on the scale increases, pain tolerance decreases, and as the score decreases, tolerance increases. The child is asked to choose the face that best expresses their emotions.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University Training and Research Hospital, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No